CLINICAL TRIAL: NCT05171660
Title: A Randomized, Open, Multicenter Phase III Clinical Trial of Combination of Sintilimab Injection (IBI308) and XELOX+Bevacizumab Compared With XELOX+Bevacizumab as 1st Line Therapy of RAS-Mutant Metastatic Colorectal Cancer
Brief Title: Combination With Sintilimab and XELOX+Bevacizumab as 1st Line Therapy in RAS-mutant Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1013
Record Dates: First submitted 2021-11-08; First posted 2021-12-29 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer Stage IV
Keywords: Colorectal Cancer Stage IV,; RAS gene mutation; Microsatellite stable
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sintilimab; Bevacizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sintilimab + XELOX + Bevacizumab (Experimental): Sintilimab + XELOX + Bevacizumab
  Interventions: Drug: Sintilimab; Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Capecitabine
- XELOX + Bevacizumab (Active Comparator): XELOX + Bevacizumab
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Sintilimab — Sintilimab Injection: 200 mg, i.v., D1, Q3W
  Arms: Sintilimab + XELOX + Bevacizumab
Drug: Bevacizumab — intravenous bevacizumab (7.5 mg/kg, day 1) in each 21-day cycle
Drug: Oxaliplatin — intravenous oxaliplatin (130 mg/m2, day 1) in each 21-day cycle
Drug: Capecitabine — oral capecitabine (1 g/m2, days 1-14) in each 21-day cycle

SUMMARY:
Sintilimab (R&D code: IBI308) is a recombinant human-derived IgG4 type PD-1 monoclonal antibody. PD-1 inhibitor combined with chemotherapy has synergistic effect to further enhance anti-tumor immunity. This study is a phase III clinical study of a three-week regimen of sintilimab combined with the XELOX+ bevacizumab for RAS-mutant metastatic colorectal cancer patients who had not received any treatment before. The purpose of this study is to explore the efficacy of sintilimab combined with XELOX + bevacizumab as first line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years old, ≤ 75 years old
2. Metastatic colorectal adenocarcinoma confirmed by histology, metastases cannot be removed
3. RAS mutation, BRAF V600E wild type, and microsatellite stable
4. ECOG 0 to 1
5. Life expectancy is at least 12 weeks
6. Hematological examination absolute neutrophil count (ANC)>1.5×109/L, hemoglobin>8g/dL and platelet>100×109/L (according to the normal value of clinical trial center)
7. Prothrombin time (PT) < 1.5 times the upper limit of normal value and normal thromboplastin time (APTT) < 1.5 times the upper limit of normal value
8. Laboratory examination, serum creatinine is less than or equal to 1.5 times the upper limit of the normal reference range (if serum creatinine is elevated, 24 hours of urine must be collected, except for 24 hours creatinine clearance > 50ml/min)
9. When there is no liver metastasis, ALT or AST is less than or equal to 2.5 times the upper limit of the normal value reference range, serum total bilirubin is less than or equal to 1.5 times the upper limit of the normal value reference range; for patients with liver metastasis, ALT or AST is less than or equal to 5 times the upper limit of the normal value reference range, serum total bilirubin is less than or equal to 3 times the upper limit of the normal value reference range
10. Women of childbearing age must be willing to use adequate contraception during study drug treatment
11. Informed consent has been signed
12. According to the definition of RECIST 1.1, the investigator determined that the patient had a measurable disease. Tumor lesions located in previous radiotherapy areas are considered measurable if they demonstrate progression.

Exclusion Criteria:

1. Active autoimmune disease requiring systemic treatment occurred in the previous 2 years.
2. Diagnosed as immunodeficiency or experimental treatment is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose. After consultation with the sponsor, the use of a physiological dose of corticosteroids may be approved.
3. Adverse events caused by anti-tumor monoclonal antibodies (mAbs) within 4 weeks prior to study day 1 or drugs received 4 weeks prior to the study have not recovered.
4. Adverse events caused by chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1, or previously received drugs, have not recovered (ie, ≤1 or reached baseline levels).

   Other malignancies that are progressing or require active treatment are known. Except for basal cell carcinoma, cutaneous squamous cell carcinoma, or cervical carcinoma in situ that have undergone radical treatment.
5. Active central nervous system (CNS) metastasis and/or cancerous meningitis are known to exist.
6. There are active infections that require systemic treatment.
7. It is possible to confuse the test results, the medical history or disease evidence, the treatment or laboratory value abnormalities that hinder the subject's full participation in the study, or the investigator believes that participating in the study is not in the best interests of the subject.
8. There are known mental or substance abuse disorders that may have an impact on compliance with test requirements.
9. Female subjects who are pregnant or lactating, or who are expected to be pregnant during the planned trial period (from 120 days after screening visits to 120 days after the last dose of study treatment, or 180 days after the last dose of study treatment), or Male subjects whose spouse is pregnant.
10. A history of infection with human immunodeficiency virus (HIV) (HIV 1/2 antibody) is known.
11. Active hepatitis B or C.
12. Live vaccines were vaccinated within 30 days of the start date of the study treatment plan.
13. RAS wild type

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival time | From randomization to the first documented disease progression, or to death from any cause, up to 2 years
  Progression-free survival is defined as the time from randomization to the first documented disease progression according to RECIST version 1.1, or to death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Objective Response Rate | From randomization to disease progression
  According to RECIST 1.1 criteria, the proportion of patients whose tumor efficacy was evaluated as CR and PR among all evaluable patients
Overall survival time | From randomization to death from any cause, up to 3 years
  Time from randomization to death from any cause
Disease control rate | From randomization to disease progression
  According to RECIST 1.1 criteria, the proportion of subjects whose tumor efficacy was evaluated as CR, PR and SD among all evaluable patients
Clinical benefit rate | From randomization to disease progression
  The proportion of patients who achieved CR PR or maintained SD for a certain period of time (6 months)
Adverse Events | From randomization to 28 days after disease progression
  Incidence of AEs (all grades), incidence of grade 1-2 AEs, incidence of grade 3-4 AEs, incidence of grade 5 AEs, treatment discontinuation rate, discontinuation rate due to adverse reactions, all subjects who used at least one study drug were included

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Xuefeng Fang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fang X, Zhong C, Weng S, Hu H, Wang J, Xiao Q, Wang J, Sun L, Xu D, Liao X, Dong C, Zhang S, Li J, Ding K, Yuan Y. Sintilimab plus bevacizumab and CapeOx (BBCAPX) on first-line treatment in patients with RAS mutant, microsatellite stable, metastatic colorectal cancer: study protocol of a randomized, open-label, multicentric study. BMC Cancer. 2023 Jul 18;23(1):676. doi: 10.1186/s12885-023-11139-z. PMID 37464378